CLINICAL TRIAL: NCT00849212
Title: A Phase II, Open-label, Ascending High-dose, add-on Study of E2007 in Patients With Refractory Partial Seizures Uncontrolled With Other Anti-epileptic Drugs (AEDs)
Brief Title: An add-on Study of E2007 in Patients With Refractory Partial Seizures Uncontrolled With Other Anti-epileptic Drugs (AEDs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-J081-231
Record Dates: First submitted 2009-02-20; First posted 2009-02-23 (Estimated); Results first posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-01

CONDITIONS: Refractory Partial Seizures
Keywords: Seizures; epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — perampanel

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E2007

INTERVENTIONS:
Drug: E2007 — The dose of E2007 will start from 2 mg and will be increased by 2 mg every week up to 12 mg (the maximum dose). The dose will be adjusted during 6 weeks (i.e., titration period). Subsequently, the dose will be fixed and maintained during 4 weeks (Maintenance period). Patients must visit study site at Weeks -4, 1, 2, 3, 4, 5, 6, 8, 10 and 14 to confirm.

SUMMARY:
The purpose of this study is to explore the maximum tolerated dose of E2007 in Japanese patients with refractory partial seizures which are uncontrolled with other anti-epileptic drugs (AEDs). Thirty patients will receive E2007 (dose escalating to the maximum of 12 mg per day). The dose of E2007 will be adjusted during 6 weeks. Subsequently, the dose will be fixed and maintained during 4 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged between 20 and 64 years old.
2. Patients diagnosed with partial seizure (including secondarily generalized seizure).
3. Patients who have at least 3 counts of partial seizures during the previous 4 weeks prior to observation start and no seizure-free for 21 days during 8 weeks before the treatment start based on medical records. Simple partial seizure without motor signs will not be counted.
4. Patients who have been treated for at least 12 weeks but confirmed to be uncontrolled with more than one standard AED for 2 years.
5. Patients treated with stable doses of up to three AEDs. Only one cytochrome

   P450 (CYP) 3A4 inducer shown below will be allowed for concomitant use:
   * Carbamazepine
   * Phenytoin
   * Phenobarbital
   * Primidone
6. Patients on stable dose of anti-depressants, anti-anxiety drugs, or mood stabilizers from before 8 weeks.

Exclusion criteria:

1. Patients with present or a history of Lennox-Gastaut syndrome.
2. Patients with present generalized seizures (e.g., absence, myoclonic).
3. Patients with a history of status epilepticus within 1 year.
4. Patients with seizure clusters where individual seizure cannot be counted within 8 weeks.
5. Patients with a history of psychogenic seizure.
6. Patients who underwent surgical operation for epilepsy within 2 years.
7. Patients using rescue benzodiazepines at least twice in a 4-week duration within 8 weeks (if 1 or 2 doses over 24-hour period considered one-time rescue).
8. Patients whose alanine aminotransferase (ALT) or aspartate aminotransferase (AST) at enrollment in observation period exceeds 1.5-fold the upper limit of normal (ULN), but those whose ALT or AST are constantly higher than ULN, they can enroll if ALT or AST remain in 3-fold the ULN.
9. Patients with significant active hematological disease; white blood cell (WBC) count </=2500/uL or neutrophil count </=1000 uL.
10. Patients on anti-psychotics or who have psychotic disorder and/or psychotic disorder(s) or unstable recurrent affective disorder(s) with a history of suicidal attempt within 2 years.
11. Patients who operate heavy equipment or drive should not be recruited into the study.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hidetaka Hiramatsu, Study Director — New Drug Development Department, Eisai Company Limited
Locations (9):
- Japan (9):
  - Kitakyushu, Fukuoka
  - Kobe, Hyōgo
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Nagasaki, Nagasaki
  - Niigata, Niigata
  - Shizuoka, Shizuoka
  - Komatsushimachō, Tokushima
  - Kodaira, Tokyo

REFERENCES:
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel: Orally administered E2007 (2, 4, 6, 8, 10, and 12 mg) once daily before bedtime (in fed administration insofar as possible). The dose started from 2 mg and up-titrated weekly in 2 mg increments up to the maximum 12 mg unless subjects met the following judgment on dose titration: 1.) If meeting titration limiting criteria, 2.) If subjects refused up-titration due to AEs, 3.) If the investigator judged it difficult to up-titrate due to AEs, or 4.) If treatment duration was less than 5 days. Total duration of treatment was 10 weeks from the initial dose.
Period: Overall Study
Arm/Group | Perampanel
Started | 30
Completed | 23
Not Completed | 7
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 2
Not completed — Miscellaneous | 1

BASELINE CHARACTERISTICS:
Arm/Group | Perampanel
Number analyzed (Participants) | 30
Age Continuous [Mean (Standard Deviation); unit: Years] — Safety analysis set
  Years | 35.4 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety analysis set: The population after excluding the following patients: a) Patients who do not meet the inclusion criteria regarding "indication," b) Patients untreated c) Patients with no evaluable data on safety
  Participants
    Female | 14
    Male | 16

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD was defined by participants. For participants who completed treatment, MTD was dose at last administration. For subjects who discontinued due to adverse event (AE), the MTD depended on the number of days within down-titration. If these criteria were not applied, the MTD was determined based on suggestions from the Tolerability and Safety Evaluation Committee.
Time Frame: 10 weeks (Titration and Maintenance Periods)
Population: Safety analysis set
Measure: Number; unit: Participants
Arm/Group | Perampanel
Number analyzed (Participants) | 30
Participants
  0 mg | 0
  2 mg | 2
  4 mg | 1
  6 mg | 6
  8 mg | 6
  10 mg | 5
  12 mg | 10

2. Secondary Outcome: Percent Change in Total Seizure Frequency Per 28 Days From Baseline (Maintenance Period) ; LOCF
Description: The percent change in seizure frequency per 28 days during the maintenance period was collected via patient diary cards. This was calculated using the last observation carried forward (LOCF) method.
Time Frame: Baseline (Day -28 to Day 0), Week 1 to Week 10
Population: Efficacy analysis set:
  Population after excluding : (a) Patients who do not meet the inclusion criteria, (b) Patients who meet the exclusion criteria which affect efficacy evaluation of E2007, (c) Patients untreated,(d) Patients with no evaluable data on efficacy,(e) Patients with <80% treatment compliance
Measure: Median (Full Range); unit: Percent change
Arm/Group | Perampanel
Number analyzed (Participants) | 27
Percent change | -35 [-100 to 312.8]

ADVERSE EVENTS:
Arm/Group | Perampanel
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 27/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=30)
Nasopharyngitis (Infections and infestations) | 5
Dizziness (Nervous system disorders) | 16
Somnolence (Nervous system disorders) | 14
Headache (Nervous system disorders) | 3
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 2
Irritability (General disorders) | 3
Malaise (General disorders) | 2
Blood creatine phosphokinase increased (Investigations) | 2
Blood glucose decreased (Investigations) | 2
Contusion (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No